CLINICAL TRIAL: NCT06084494
Title: An Experimental Investigation of Physiological Responses in Semiprofessional Athletes: Comparing the Impact of Climatic Conditions, Physical Activity, and Gender
Brief Title: Validation of Heat Stress Limit Values for the Athletic Performance
Acronym: HSL-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Punjab (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Muhammad Salman Butt, Clinical Trial Coordinator, University of the Punjab
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: VEN 99 -11
Record Dates: First submitted 2023-08-02; First posted 2023-10-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Physiological Stress; Heat Stress; Sports Injury; Heat Stress, Exertional
Keywords: Heat Stress; Physiological Responses; WBGT; PHS
MeSH Terms: conditions — Heat Stress Disorders; Athletic Injuries

STUDY DESIGN:
Intervention Model Description: A wet Bulb Globe temperature (WBGT) level of 28 °C was simulated, and the temperature within the climatic chamber was set at 40 °C and 31 °C at relative humidity levels of 20% and 70%, respectively. Four test conditions were designed and subjects ran at 8 km/h and walked at 5 km/h for up to 70 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Condition 1 (Experimental): Variable Test Condition 1 WBGT 28 °C Clothing High Visibility Air Temperature 40 °C RH % 20 % Vapor Pressure 2.3 kPa Walking Speed 5 km/h Time 70 min
  Interventions: Diagnostic Test: analytical determination and interpretation of heat stress using calculation of the Predicted Heat Strain and Wet Bulb Globe Temperature
- Test Condition 2 (Experimental): Variable Test Condition 2 WBGT 28 °C Clothing High Visibility Air Temperature 40 °C RH % 20 % Vapor Pressure 2.3 kPa Walking Speed 8 km/h Time 70 min
  Interventions: Diagnostic Test: analytical determination and interpretation of heat stress using calculation of the Predicted Heat Strain and Wet Bulb Globe Temperature
- Test Condition 3 (Experimental): Variable Test Condition 3 WBGT 28 °C Clothing High Visibility Air Temperature 31 °C RH % 70 % Vapor Pressure 3.1 kPa Walking Speed 5 km/h Time 70 min
  Interventions: Diagnostic Test: analytical determination and interpretation of heat stress using calculation of the Predicted Heat Strain and Wet Bulb Globe Temperature
- Test Condition 4 (Experimental): Variable Test Condition 4 WBGT 28 °C Clothing High Visibility Air Temperature 31 °C RH % 70 % Vapor Pressure 3.1 kPa Walking Speed 8 km/h Time 70 min
  Interventions: Diagnostic Test: analytical determination and interpretation of heat stress using calculation of the Predicted Heat Strain and Wet Bulb Globe Temperature

INTERVENTIONS:
Diagnostic Test: analytical determination and interpretation of heat stress using calculation of the Predicted Heat Strain and Wet Bulb Globe Temperature — The temperature inside the climatic chamber was set at 40 C and 31 C at a relative humidity of 20 % and 70 % respectively to count for a WBGT level of 28 C. The subject does walk at 5 km/h and jog at 8 km/h under these conditions for up to 70 minutes. The test includes the measurement of the height and weight of the subjects, heart rate, oxygen consumption, body weight loss (sweat evaporation), skin temperature, and core body temperature under hot environmental conditions. Subjective responses will also be recorded. WBGT was recorded after every ten minutes by heat stress meter and Bruel Kjaer.

SUMMARY:
Three male and three female semi-professional athletes, ranging in age from 22 to 27, participated in a study that was done at Lund University in Sweden to examine their physiological responses. The temperature and relative humidity were adjusted at 40 degrees Celsius for hot, dry conditions and 31 degrees Celsius for hot, wet conditions, respectively. The participants were instructed to engage in physical activity on a treadmill within the chamber for 70 minutes, or until participants were able to continue their exercise without difficulty within the allotted period. Participants were instructed to walk (5 kph) and run (8 kph). Participants pulse rate, breathing rate, oxygen consumption, and subjective reactions were all recorded.

On the basis of the Wet Bulb Globe Temperature (WBGT), a heat stress index, the American College of Sports Medicine has made certain suggestions. The technique used to determine the temperature on a Celsius scale took into account the influences of relative humidity, air temperature, wind, and direct sunlight radiation. The American College of Sports Medicine advises delaying athletic competition when the WBGT is above 28 degrees. In the climate control chamber, the trials were carried out in high-risk circumstances (28 degrees Celsius WBGT). According to the study's findings, exercise is influenced by weather, and as air temperature rises, so do the intensity of exertion and thermal feeling.

DETAILED DESCRIPTION:
Methodology Experimental research design Study Duration 6 months Study Centres Thermal Environment Laboratory, Department of Design Sciences, Faculty of Engineering (LTH), Lund University Main Objectives Objective 1: To examine the physiological responses (skin temperature, core body temperature, body temperature, heart rate, and oxygen uptake) of semi-professional athletes during physical activity in different climatic conditions (hot wet and hot dry) Objective 2: To compare the effects of physical activity intensity (5 km/hr and 8 km/hr) on the physiological responses of semi-professional athletes under varying climatic conditions.

Objective 3: To investigate the influence of gender on the physiological responses of semi-professional athletes during physical activity in different climatic conditions.

Objective 4: To assess the suitability of the Physiological Heat Strain (PHS) and Wet Bulb Globe Temperature (WBGT) index for evaluating heat stress in sports settings based on the findings from semi-professional athletes.

No. of Participants Six semiprofessional athletes including three males and three females with a mean age of (24.7 ± 2.1 years) and a body surface area mean of (1.8 ± 0.2 m2) participated in this study.

Main Eligibility Criteria Key factors to consider when defining semiprofessionals include participation in regional competition level, receiving monetary compensation for their sports participation, participating in sports activity in the last six years, and skill level. These athletes typically demonstrate a higher level of skill and performance than recreational or amateur participants.

ELIGIBILITY:
Inclusion Criteria

* Semiprofessional aged 22-27 years of both genders.
* Body surface area between 1.5 to 2.5 m2
* Semiprofessional participating in regional competition level, receive monetary compensation for their sports participation, participating in sports activity in the last six year, and skill level.
* Semiprofessional demonstrating a higher level of skill and performance than recreational or amateur participants .

Exclusion Criteria

* Subjects should not have any known heart disease or circulatory disorder.
* No known respiratory disease or heat allergy.
* No habitual smoker or drug user.

Ages: 22 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Six semiprofessional athletes including three males and three females with a mean age of (24.7 ± 2.1 years) and a body surface area mean of (1.8 ± 0.2 m2) participated in this study.
Enrollment: 6 (Actual)
Dates: Start 2012-10-21 (Actual); Primary Completion 2013-02-01 (Actual); Study Completion 2013-12-30 (Actual)

PRIMARY OUTCOMES:
Physiological Response | 70 minutes
  Rate of change of skin temperature (Tsk) of semi-professional athletes during walking 5km/hr and Jogging 8km/hr for 70 minutes in hot wet (Ta 40 C & 70% RH) and hot dry (Ta 31C & 20% RH) test conditions.
Physiological Response | 70 minutes
  Rate of change of core body temperature (Tcore) of semi-professional athletes during walking 5km/hr and Jogging 8km/hr for 70 minutes in hot wet (Ta 40 C & 70% RH) and hot dry (Ta 31 C & 20% RH) test conditions.
Physiological Response | 70 minutes
  Rate of change of Heart Rate (HR bpm) of semi-professional athletes during walking 5km/hr and Jogging 8km/hr for 70 minutes in hot wet (Ta 40 C & 70% RH) and hot dry (Ta 31 C & 20% RH) test conditions.
Physiological Response | 70 minutes
  Consumption of oxygen (VO2 Max ml/min/kg) of semi-professional athletes during walking 5km/hr and Jogging 8km/hr for 70 minutes in hot wet (Ta 40 C & 70% RH) and hot dry (Ta 31 C & 20% RH) test conditions.

SECONDARY OUTCOMES:
Gender-Based Physiological Responses | 70 minutes
  Gender-based comparison of the change in core body temperature of semi-professional athletes while performing various physical activities at 28 C WBGT
Heat Stress Indices | 70 minutes
  Comparison of Physiological Heat Strain (PHS) and Wet Bulb Globe Temperature (WBGT) index for evaluating heat stress in sports settings based on the core body temperature responses from semi-professional athletes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health, University of the Punjab, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-08-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT06084494/Prot_SAP_ICF_000.pdf